CLINICAL TRIAL: NCT02592447
Title: Preliminary Evaluation of an Internet-Assisted Cognitive Behavioral Intervention for Targeted Therapy Fatigue
Brief Title: Cognitive Behavioral Intervention for Targeted Therapy Fatigue (CBT-TTF) Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-18365; R21CA191594 (NIH)
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: CML; chronic phase CML; leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase; Leukemia | interventions — Therapeutics; Behavior Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavior Therapy (CBT) (Experimental): Cognitive Behavior Therapy for Targeted Therapy-related Fatigue (CBT-TTF) to help manage fatigue via FaceTime on an iPad, which will be provided to participants. Participants will meet with a trained therapist who will outline their therapy plan and will be taught how to use the iPad for upcoming therapy sessions.
  Interventions: Other: Therapy for Targeted Therapy-related Fatigue (TTF)
- Wait-List Control Condition (WLC) (Other): Wait-List Control Condition (WLC) group will not receive therapy sessions and will continue usual care with their providers. This group will be offered the same cognitive behavior therapy as the group receiving the CBT-TTF intervention, after the 18 week study period.
  Interventions: Other: Wait-List Control Condition (WLC)

INTERVENTIONS:
Other: Therapy for Targeted Therapy-related Fatigue (TTF) — Cognitive Behavior Therapy for Targeted Therapy-related Fatigue (CBT-TTF) group will receive cognitive behavior therapy to help manage fatigue via FaceTime on an iPad, which will be provided to participants. Participants will meet with a trained therapist who will outline their therapy plan and will be taught how to use the iPad for upcoming therapy sessions. The sessions will initially be held weekly, but the therapist may schedule sessions at 1-, 2-, or 3-week intervals during the 18 week study period. The final session will be conducted either in-person at Moffitt or via FaceTime.
  Other Names: behavioral therapy
  Arms: Cognitive Behavior Therapy (CBT)
Other: Wait-List Control Condition (WLC) — Participants randomized to Wait-List Control Condition will continue to receive care under direction of their Moffitt Cancer Center (MCC) physician. Physicians will be informed by email of patients' participation on the basis of elevated fatigue and their randomization to WLC. Chart review and a patient self-report form will be used at baseline and follow-up assessments to determine what, if any, services or interventions participants received in the preceding 18 weeks that might address fatigue.
  Other Names: standard of care; SOC
  Arms: Wait-List Control Condition (WLC)

SUMMARY:
The purpose of this study is to evaluate Cognitive Behavioral Intervention for Targeted Therapy Fatigue (CBT-TTF) with fatigued chronic myelogenous leukemia (CML) patients on tyrosine kinase inhibitors (TKIs) for feasibility, acceptability and potential efficacy relative to usual care only in a small-scale randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* able to speak/read English
* diagnosed with chronic phase CML
* not have been treated for other cancer (except non-melanoma skin cancer) in the past 5 years
* be under the care of a Moffitt Cancer Center (MCC) physician
* be on a stable dose of the same oral TKI for >= 3 months
* new onset or worsening of fatigue since starting TKI
* report moderate-severe fatigue in past week (FSI average rating >= 4 of 0-10)
* have no clinical history of disease (e.g., multiple sclerosis, fibromyalgia) that could account for their fatigue presentation

Exclusion Criteria:

* scheduled to discontinue their TKI under medical supervision within the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Jim, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Oswald LB, Hyland KA, Eisel SL, Hoogland AI, Knoop H, Nelson AM, Pinilla-Ibarz J, Sweet K, Jacobsen PB, Jim HSL. Correlates of fatigue severity in patients with chronic myeloid leukemia treated with targeted therapy. Support Care Cancer. 2022 Jan;30(1):87-94. doi: 10.1007/s00520-021-06408-1. Epub 2021 Jul 7. PMID 34231041
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 48 consented, 4 never completed questionnaires.
Period: Overall Study
Arm/Group | Cognitive Behavior Therapy (CBT) | Wait-List Control Condition (WLC)
Started | 29 | 15
Completed | 27 | 14
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Ineligible after randomization | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavior Therapy (CBT) | Wait-List Control Condition (WLC) | Total
Number analyzed (Participants) | 29 | 15 | 44
Age, Continuous [Mean (Full Range); unit: years] | 53 [29 to 82] | 60 [39 to 78] | 55 [29 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 15 | 8 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 26 | 12 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Fatigue Scores - Change From Baseline Per Scoring Category
Description: Baseline versus follow-up fatigue will be assessed with the Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-Fatigue) v.4, a 13-item self-report measure yielding total score with demonstrated reliability, validity, sensitivity to change and an identified Minimally Clinically Important Difference (MID). The fatigue subscale consists of 13 items asking about fatigue in the past 7 days. Items are summed to produce a score ranging from 0-52 with lower scores indicating greater fatigue. A difference of 3 points on the fatigue subscale indicates a clinically-important difference.
Time Frame: Baseline and at 18 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavior Therapy (CBT) | Wait-List Control Condition (WLC)
Number analyzed (Participants) | 27 | 14
score on a scale
  Fatigue score at baseline | 28.03 (6.92) | 24.53 (7.05)
  Fatigue score at 18 weeks | 15.7 (8.69) | 24.7 (8.18)

2. Secondary Outcome: Self-reported Quality of Life (QoL) Scores - Change From Baseline Per Scoring Category
Description: Baseline versus follow-up quality of life will be assessed with the Functional Assessment of Cancer Therapy General Scale (FACT-G) v.4, a 27-item measure yielding total score and scores for physical, social/family, emotional, and functional well-being of demonstrated reliability, validity, and sensitivity to change. FACT-G consists of 4 subscales: physical well-being (PWB), functional well-being (FWB), emotional well-being (EWB) and social well-being (SWB). Scores on the four subscales are summed to produce a total score ranging from 0 to 108 with higher scores indicating better quality of life.
Time Frame: Baseline and at 18 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavior Therapy (CBT) | Wait-List Control Condition (WLC)
Number analyzed (Participants) | 27 | 14
score on a scale
  Quality of Life Score at Baseline | 64.04 (15.05) | 63.83 (14.44)
  Quality of Life Score at 18 weeks | 84.25 (15.37) | 68.22 (10.59)

ADVERSE EVENTS:
Description: All Cause Mortality, Serious and Other Adverse Events were not monitored/assessed
Arm/Group | Cognitive Behavior Therapy (CBT) | Wait-List Control Condition (WLC)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT02592447/Prot_SAP_000.pdf